CLINICAL TRIAL: NCT01700933
Title: Dose-response: Exercise Therapy on Hip Osteoarthritis, a Pilot Study
Brief Title: Dose-response: Exercise Therapy on Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DROAPS1
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis, Hip
Keywords: Exercise therapy
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dosage-group (Active Comparator)
  Interventions: Other: High-Dosage Exercise Therapy
- Low-dosage-group (Active Comparator)
  Interventions: Other: Low-Dosage Exercise Therapy

INTERVENTIONS:
Other: High-Dosage Exercise Therapy — Structure of the exercise program done three times per week, for eight weeks:
  5-10 minutes of global exercise (cycling, walking on treadmill etc.) Four local exercises (3 series of 30 repetitions) 5-10 minutes of global exercise (cycling, walking on treadmill etc.) Four local exercises (3 series of 30 repetitions) 5-10 minutes of global exercise (cycling, walking on treadmill etc.)
  Arms: High-dosage-group
Other: Low-Dosage Exercise Therapy — Structure of the exercise program done three times per week, for eight weeks:
  5-10 minutes of global exercise (cycling, walking on treadmill etc.) Four local exercises (3 series of 10 repetitions) 5-10 minutes of global exercise (cycling, walking on treadmill etc.) Four local exercises (3 series of 10 repetitions) 5-10 minutes of global exercise (cycling, walking on treadmill etc.)
  Arms: Low-dosage-group

SUMMARY:
Osteoarthritis is a common disease that causes muscle weakness, stiffness and instability. The disease reduces the opportunities for an active lifestyle. Exercise Therapy provides a well-documented effect on pain and function in patients with osteoarthritis of the hip. It is sought an optimal dose of exercise, in which this study will help to investigate.

We hypothesize that an exercise program designed to have a high number of repetitions will benefit the outcome of the training in a more positive way than a low-repetition based program.

ELIGIBILITY:
Inclusion Criteria:

* At least three month since debut of the disease
* Age above 45 years
* Ability to complete the intervention

Exclusion Criteria:

* Pain above 4 on VAS during gait
* Pregnancy
* Autoimmune disease
* Cardiovascular disease
* Respiratory disease
* Metabolic disease
* Neurological signs
* Planned hip-replacement surgery within the next year
* Received exercise therapy within the last 3 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
WOMAC Index of Osteoarthritis (questionnaire) | 0 weeks, 8 weeks, 6 months postinterventional
  WOMAC Index of Osteoarthritis (questionnaire)

SECONDARY OUTCOMES:
HAD questionnaire | 0 weeks, 8 weeks, 6 months postinterventional
Tampa Scale for Kinesiophobia | 0 weeks, 8 weeks, 6 months postinterventional
Squats | 0 weeks, 8 weeks, 6 months postinterventional
  Number of squats completed in 30 seconds.
Stairs | 0 weeks, 8 weeks, 6 months postinterventional
  Time used to walk up and down 12 steps.

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Østerås, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Fysioterapitjenesten i Ørsta, Ørsta, Norway

REFERENCES:
- [Result] Osteras H, Paulsberg F, Olsen SE, Osteras B, Torstensen TA. Effects of medical exercise therapy in patients with hip osteoarthritis: A randomized controlled trial with six months follow-up. A pilot study. J Bodyw Mov Ther. 2017 Apr;21(2):284-289. doi: 10.1016/j.jbmt.2016.06.016. Epub 2016 Jul 5. PMID 28532870